CLINICAL TRIAL: NCT00272753
Title: A Randomized Double Blind Comparison Between Single Doses of Symbicort Turbuhaler (Budesonide/Formoterol Combination), Formoterol, Salbutamol and Placebo in Repeated AMP-challenges in Patients With Mild - to Moderate Asthma. Investigating the Supplementary Value of the Budesonide Component Within Symbicort When Tested in a Model of Slow Onset Acute Asthma
Brief Title: Effect of Budesonide / Formoterol Combination in Repeated AMP Provocations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BN-00S-0022
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: budesonide/formoterol Turbuhaler
  Other Names: Symbicort
Drug: formoterol Turbuhaler
Drug: salbutamol

SUMMARY:
The aim is to study whether the budesonide component within the budesonide/ formoterol combination inhaler has additive value in a model of "slow onset acute asthma" , namely three AMP provocation tests performed on one day

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosis according to ATS criteria,
* lung function (FEV1) above 60% of predicted,
* AMP-PC20 below 160 mg/ml with a documented fall in FEV1 of 30% in this provocation test

Exclusion Criteria:

* having smoked > 10 Pack-years,
* hypersensitivity to one of the study drugs,
* significant co-morbidity, pregnancy or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
The decrease in lung function (FEV1) after the third AMP provocation test.

SECONDARY OUTCOMES:
Decrease in lung function (FEV1) after the second AMP provocation test,
lung function and Borg Score over the test day,
increase in FEV1 at three minutes after study drug inhalation,
time course of recovery from the AMP-induced decrease in lung function

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Groningen

REFERENCES:
- [Derived] Aalbers R, Boorsma M, van der Woude HJ, Jonkers RE. Protective effect of budesonide/formoterol compared with formoterol, salbutamol and placebo on repeated provocations with inhaled AMP in patients with asthma: a randomised, double-blind, cross-over study. Respir Res. 2010 May 28;11(1):66. doi: 10.1186/1465-9921-11-66. PMID 20509942